CLINICAL TRIAL: NCT01546792
Title: Effects of a Lifestyle Intervention on Quality of Life, Weight Loss and Cardiovascular Risk in Patients With Obstructive Sleep Apnoea Established on Continuous Positive Airway Pressure
Brief Title: Lifestyle Intervention in Obstructive Sleep Apnoea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other)
Responsible Party: Principal Investigator, Garry Tew, Senior Research Fellow, Sheffield Teaching Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STH15488
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Obstructive Sleep Apnoea; Obesity
Keywords: exercise; diet; lifestyle; sleep apnoea; obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity; Motor Activity; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care control (No Intervention): Leaflet on exercise and diet
- Lifestyle intervention (Experimental): Exercise training (mixture of supervised and non-supervised) Dietary advice Behaviour change counselling (physical activity, diet)
  Interventions: Behavioral: Combined lifestyle intervention

INTERVENTIONS:
Behavioral: Combined lifestyle intervention — Exercise training, dietary advice, behaviour change counselling
  Arms: Lifestyle intervention

SUMMARY:
Obstructive sleep apnoea/hypopnoea syndrome (OSAHS) is a common disorder characterised by interrupted breathing while sleeping. It is associated with cardiovascular problems such as high blood pressure, heart attack and stroke. Furthermore, most patients with OSAHS are overweight and have impaired quality of life. Lifestyle interventions incorporating exercise training, dietary advice and behaviour change have been shown to elicit favourable changes in quality of life, body mass/composition and cardiovascular risk in a range of patient groups. However, no study has investigated the impact of lifestyle modification on such health outcomes in patients with OSAHS. This study will address this issue by investigating the effects of a lifestyle intervention on quality of life, body mass/composition and cardiovascular risk in patients with OSAHS. A total of 60 volunteers will be recruited and randomly allocated to one of the two groups. Patients in the intervention group will be offered a 12-week individualised lifestyle programme consisting of supervised exercise training, dietary advice and behaviour change counselling. Patients in the control group will receive an educational booklet detailing healthy eating and exercise guidelines but no supervised or structured intervention. The results of this study will inform the design of a larger, multi-centre randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* obstructive sleep apnoea patients who have been receiving CPAP therapy for at least 6 months and are known to be adherent to the treatment (>75% nightly use per week)
* clinically obese (body mass index >30)
* age 18-85 years
* able to undertake exercise testing and training

Exclusion Criteria:

* patients with any contraindications to exercise (e.g. severe hypertension, unstable arrhythmias, severe musculoskeletal injuries)
* unable to undertake the requirements of the study
* non-English speaking
* already undertaking >30 min exercise >3 times per week
* non-compliant with CPAP
* body mass index <30
* unable to provide written informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Body mass | 25 weeks
Incremental shuttle walk performance | 25 weeks

SECONDARY OUTCOMES:
Quality of life (EQ-5D and EQ-VAS) | 13 and 25 weeks
Body fat percentage | 13 and 25 weeks
Resting blood pressure | 13 and 25 weeks
Blood markers (glucose, insulin, lipids, CRP) | 13 and 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bianchi, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Centre for Sport and Exercise Science, Sheffield Hallam University, Sheffield, South Yorkshire
  - Pulmonary Function Unit, Northern General Hospital, Sheffield, South Yorkshire

REFERENCES:
- [Derived] Moss J, Tew GA, Copeland RJ, Stout M, Billings CG, Saxton JM, Winter EM, Bianchi SM. Effects of a pragmatic lifestyle intervention for reducing body mass in obese adults with obstructive sleep apnoea: a randomised controlled trial. Biomed Res Int. 2014;2014:102164. doi: 10.1155/2014/102164. Epub 2014 Jul 21. PMID 25136550